CLINICAL TRIAL: NCT03300401
Title: The Role of Quantitative Contrast-Enhanced Ultrasound in Yttrium-90 (90Y) Radioembolization of Hepatocellular Carcinoma
Brief Title: Contrast-Enhanced Ultrasound in Diagnosing Patients With Liver Cancer Undergoing Yttrium-90 Radioembolization
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Accrual issue
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 3L-17-3; NCI-2017-01422 (Registry Identifier: Registry ID: CTRP (Clinical Trial Reporting Program)); 3L-17-3 (Other: USC/Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2017-09-27; First posted 2017-10-03 (Actual); Last update posted 2019-05-16 (Actual); Status verified 2019-05

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — perflutren; Positron-Emission Tomography; Tomography, X-Ray Computed; Yttrium-90

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Diagnostic (CEUS) (Experimental): Patients receive perflutren or sulfur hexafluoride lipid microspheres and undergo CEUS at baseline, 2 and 4 weeks, and 3 and 6 months. Patients also undergo PET/CT after standard of care 90Y radioembolization at baseline.
  Interventions: Drug: Perflutren Lipid Microspheres; Drug: Sulfur Hexafluoride Lipid Microspheres; Device: Dynamic Contrast-Enhanced Ultrasound Imaging; Device: Positron Emission Tomography; Device: Computed Tomography; Biological: Yttrium-90 (90Y)

INTERVENTIONS:
Drug: Perflutren Lipid Microspheres — Receive intravenous injection just prior to ultrasound
  Other Names: Definity
Drug: Sulfur Hexafluoride Lipid Microspheres — Receive intravenous injection just prior to ultrasound
  Other Names: Lumason
Device: Dynamic Contrast-Enhanced Ultrasound Imaging — Undergo Contrast-Enhanced Ultrasound Imaging
  Other Names: Contrast-Enhanced Ultrasound Imaging
Device: Positron Emission Tomography — Undergo PET/CT
Device: Computed Tomography — Undergo CT scan
  Other Names: Computerized Axial Tomography
Biological: Yttrium-90 (90Y) — Given IV
  Other Names: 90Y microsphere

SUMMARY:
This pilot clinical trial studies how well contrast-enhanced ultrasound in diagnosing patients with liver cancer who are undergoing Yttrium-90 radioembolization. Contrast-enhanced ultrasound may provide detailed imaging of the tumor arteries after the injection of a contrast-agent consisting of microbubbles, and may predict how much Yttrium-90 will deposit in the tumor.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Investigate the relationship between hepatocellular carcinoma (HCC) tumor perfusion on pre-procedural contrast-enhanced ultrasound (CEUS) time intensity curve (TIC) and post-procedural Yttrium-90 (90Y) microsphere distribution after 90Y radioembolization (RE).

SECONDARY OBJECTIVES:

I. Study the potential of serial CEUS TIC examinations as a marker of tumor treatment response as assessed at 20 - 24 week computed tomography (CT) follow-up.

OUTLINE:

Patients receive perflutren or sulfur hexafluoride lipid microspheres and undergo CEUS at baseline, 2 and 4 weeks, and 3 and 6 months. Patients also undergo positron emission tomography/computed tomography (PET/CT) after standard of care 90Y radioembolization at baseline.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for 90Y radioembolization for HCC as part of their standard of care

Exclusion Criteria:

* Patients who have already received tumor treatment (either systemic or loco-regional such as previous Y90RE, microwave or radiofrequency [RF] ablation or transarterial chemoembolization [TACE])
* Pregnant or nursing
* Known cardiac shunt
* Known pulmonary hypertension
* History of hypersensitivity to Definity (perflutren lipid microsphere) or Lumason
* History of hypersensitivity to iodinated contrast agent
* Cannot consent for himself or herself

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-11-07 (Actual); Primary Completion 2019-11-07 (Estimated); Study Completion 2020-11-07 (Estimated)

PRIMARY OUTCOMES:
Local tumor response to therapy | Up to 24 weeks
  Will be assessed by modified Response Evaluation Criteria in Solid Tumors criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Harshawn Malhi, MD, Principal Investigator — University of Southern California
Locations (1):
- USC/Norris Comprehensive Cancer Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided